CLINICAL TRIAL: NCT02218372
Title: A Phase 3, Multicenter, Investigator-blind, Randomized, Parallel Group Study to Investigate the Safety and Efficacy of Fidaxomicin Oral Suspension or Tablets Taken q12h, and Vancomycin Oral Liquid or Capsules Taken q6h, for 10 Days in Pediatric Subjects With Clostridium Difficile-associated Diarrhea
Brief Title: A Study to Investigate the Safety and Efficacy of Fidaxomicin (Oral Suspension or Tablets) and Vancomycin (Oral Liquid or Capsules) in Pediatric Subjects With Clostridium Difficile-associated Diarrhea (CDAD)
Acronym: SUNSHINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2819-CL-0202; 2013-000508-40 (EudraCT Number); SUNSHINE (Other: Acronym)
Record Dates: First submitted 2014-08-11; First posted 2014-08-18 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Clostridium Difficile-associated Diarrhea (CDAD)
Keywords: Clostridium difficile-associated Diarrhea (CDAD); vancomycin; Clostridium difficile infection; fidaxomicin
MeSH Terms: conditions — Clostridium Infections | interventions — Fidaxomicin; Vancomycin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fidaxomicin (Experimental): Participants from birth to < 6 years of age received weight based doses of fidaxomicin oral suspension (32 mg/kg/day with a maximum dose of 400 mg/day divided in 2 doses) 2 times daily for 10 days. Participants aged ≥ 6 years to < 18 years of age received a 200 mg fidaxomicin tablet 2 times daily for 10 days.
  Interventions: Drug: Fidaxomicin oral suspension; Drug: Fidaxomicin tablets
- Vancomycin (Active Comparator): Participants from birth to < 6 years of age received weight based doses of vancomycin oral liquid (40 mg/kg/day with a maximum dose of 500 mg/day divided in 4 doses) 4 times daily for 10 days. Participants aged ≥ 6 years to < 18 years of age received a 125 mg vancomycin capsule 4 times daily for 10 days.
  Interventions: Drug: Vancomycin oral liquid; Drug: Vancomycin capsules

INTERVENTIONS:
Drug: Fidaxomicin oral suspension — Participants from birth to < 6 years of age received weight based doses of fidaxomicin oral suspension (32 mg/kg/day with a maximum dose of 400 mg/day divided in 2 doses) 2 times daily for 10 days.
  Other Names: Dificid; Dificlir
  Arms: Fidaxomicin
Drug: Fidaxomicin tablets — Participants aged ≥ 6 years to < 18 years of age received a 200 mg fidaxomicin tablet 2 times daily for 10 days.
  Other Names: Dificlir; Dificid
  Arms: Fidaxomicin
Drug: Vancomycin oral liquid — Participants from birth to < 6 years of age received weight based doses of vancomycin oral liquid (40 mg/kg/day with a maximum dose of 500 mg/day divided in 4 doses) 4 times daily for 10 days.
  Arms: Vancomycin
Drug: Vancomycin capsules — Participants aged ≥ 6 years to < 18 years of age received a 125 mg vancomycin capsule 4 times daily for 10 days.
  Arms: Vancomycin

SUMMARY:
The purpose of this study was to investigate the clinical response to fidaxomicin oral suspension or tablets and vancomycin oral liquid or capsules in pediatric participants with Clostridium difficile-associated diarrhea (CDAD). It also investigated the recurrence/sustained clinical response to and safety of fidaxomicin and vancomycin, as well as acceptance of the fidaxomicin oral suspension formulation.

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with CDAD according to local diagnostic criteria. As a minimum there must be positive detection, within 72 hours prior to randomization, of either toxin A and/or toxin B in stool or positive detection of toxigenic C. difficile in stool and:

  * Subject from Birth to < 2 years: watery diarrhea in the 24 hours prior to screening.
  * Subject ≥ 2 years to < 18 years: ≥ 3 unformed bowel movements in the 24 hours prior to screening.
  * Male and female subjects aged from birth to < 18 years: Note that in the United States of America subjects can only be included if aged ≥ 6 months to < 18 years.
* For subjects < 5 years: Negative rotavirus test.
* Female subject of childbearing potential:

  * must have a negative urine pregnancy test at Screening, and
  * must abstain from sexual activity for the duration of the study, or
  * must use two forms of birth control (at least one of which must be a barrier method) starting at Screening and throughout the study period and for 28 days after the final study drug administration.
* Female subject must not be breastfeeding at Screening or during the study period, and for 28 days after the final study drug administration.
* Female subject must not donate ova starting at Screening and throughout the study period, and for 28 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while in the study (with the exception of studies as described in exclusion criteria below).

Exclusion Criteria:

* Concurrent use of metronidazole, oral vancomycin or any other antibiotic treatments for CDAD. If the investigator feels the clinical imperative is to begin treatment before knowing the laboratory result for toxigenic C. difficile, up to four doses but no more than 24 hours of treatment with metronidazole, oral vancomycin or any other effective treatment for CDAD are allowed.
* Subject has pseudomembranous colitis, fulminant colitis, toxic megacolon or ileus.
* Subject has a history of inflammatory bowel disease (e.g., ulcerative colitis or Crohn's disease etc.).
* Subject has diarrhea caused by an agent other than C. difficile (e.g. infections, infestations, drugs etc.).
* Subject has known hypersensitivity to fidaxomicin, vancomycin or their excipients or to teicoplanin.
* Subject has received an investigational therapy within 28 days, prior to Screening, with the exception of studies with primary treatment for cancer without novel Investigational Medicinal Product (IMP) and which do not affect the assessment of diarrhea.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2015-01-09 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Research Physician, Study Director — Astellas Pharma Europe B.V.
Locations (44):
- United States (14):
  - Site US10015, Orange, California
  - Site US10010, Chicago, Illinois
  - Site US10004, Indianapolis, Indiana
  - Site US10025, Louisville, Kentucky
  - Site US10032, Kansas City, Missouri
  - Site US10030, Omaha, Nebraska
  - Site US10008, Stony Brook, New York
  - Site US10028, Chapel Hill, North Carolina
  - Site US10027, Cincinnati, Ohio
  - Site US10014, Toledo, Ohio
  - Site US10034, Johnson City, Tennessee
  - Site US10022, Memphis, Tennessee
  - Site US10038, Fort Worth, Texas
  - Site US10037, Salt Lake City, Utah
- Belgium (3):
  - Site BE32001, Brussels, Flemish Brabant
  - Site BE32003, Ghent
  - Site BE32002, Liège
- Site CA15003, Oshawa, Ontario, Canada
- France (5):
  - Site FR33002, La Tronche
  - Site FR33001, Nice
  - Site FR33007, Nice
  - Site FR33005, Paris
  - Site FR33008, Strasbourg
- Germany (6):
  - Site DE49010, Essen
  - Site DE49002, Frankfurt Am M.
  - Site DE49006, Freiburg im Breisgau
  - Site DE49004, Mainz
  - Site DE49001, Münster
  - Site DE49003, Saint Augustin
- Hungary (2):
  - Site HU36006, Budapest
  - Site HU36004, Szeged
- Italy (2):
  - Site IT39004, Milan
  - Site IT39001, Roma
- Poland (6):
  - Site PL48002, Warsaw, Masovian Voivodeship
  - Site PL48012, Bialystok
  - Site PL48007, Bydgoszcz
  - Site PL48004, Dębica
  - Site PL48014, Rzeszów
  - Site PL48006, Tarnów
- Site RO40005, Bucharest, Romania
- Spain (4):
  - Site ES34002, Barcelona
  - Site ES34007, Madrid
  - Site ES34004, Madrid
  - Site ES34003, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Wolf J, Kalocsai K, Fortuny C, Lazar S, Bosis S, Korczowski B, Petit A, Bradford D, Croos-Dabrera R, Incera E, Melis J, van Maanen R. Safety and Efficacy of Fidaxomicin and Vancomycin in Children and Adolescents with Clostridioides (Clostridium) difficile Infection: A Phase 3, Multicenter, Randomized, Single-blind Clinical Trial (SUNSHINE). Clin Infect Dis. 2020 Dec 17;71(10):2581-2588. doi: 10.1093/cid/ciz1149. PMID 31773143
- [Derived] Borali E, De Giacomo C. Clostridium Difficile Infection in Children: A Review. J Pediatr Gastroenterol Nutr. 2016 Dec;63(6):e130-e140. doi: 10.1097/MPG.0000000000001264. PMID 27182626
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=362

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric participants with clostridium difficile-associated diarrhea (CDAD) were enrolled in this multicenter study.
Pre-assignment Details: Eligible participants who met inclusion criteria and none of the exclusion criteria were enrolled, 159 participants were assessed for eligibility of whom 148 were randomized. Participants were randomized to either fidaxomicin or vancomycin in a 2:1 ratio, stratified by age group.
Period: Overall Study
Arm/Group | Fidaxomicin | Vancomycin
Started | 100 | 48
Treated | 98 | 44
Completed | 95 | 42
Not Completed | 5 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Miscellaneous | 2 | 1
Not completed — Randomized but did not receive treatment | 2 | 3
Not completed — Withdrawal by Parent/Guardian | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis set consisted of the Intent-to-treat (ITT) population. The ITT analysis set consisted of all randomized participants, irrespective of a participant having received a study drug (fidaxomicin or vancomycin) or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fidaxomicin | Vancomycin | Total
Number analyzed (Participants) | 100 | 48 | 148
Age, Continuous [Mean (Standard Deviation); unit: months] | 79.7 (61.8) | 77.5 (59.2) | 79 (60.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 21 | 62
  Male | 59 | 27 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 83 | 36 | 119
  Black or African American | 6 | 5 | 11
  Asian | 2 | 0 | 2
  Other | 4 | 1 | 5
  Missing | 5 | 6 | 11
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 5 | 17
  Not Hispanic or Latino | 82 | 37 | 119
  Missing | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Clinical Response (CCR) at End of Treatment (EOT) +2 Days
Description: Initial clinical response (ICR) for ages from birth to < 2 years was defined as absence of watery diarrhea for 2 consecutive treatment days, remaining well until study drug discontinuation. ICR for ages ≥ 2 years to < 18 years was defined as improvement in number and character of bowel movements as determined by < 3 unformed bowel movements (UBMs) per day for 2 consecutive treatment days, remaining well until study drug discontinuation. CCR was defined for both age groups as not requiring further CDAD therapy within 2 days after study drug completion, and was reported with a positive (Yes) or negative (No) outcome. Resolution of diarrhea was assessed during interviews of participant/parent/legal guardian, supplemented by review of personal records (if hospitalized) and checked for presence of watery diarrhea (ages from birth to < 2 years) or number of UBMs (for ages ≥ 2 years to < 18 years).
Time Frame: Up to day 12
Population: The analysis population consisted of the full analysis set (FAS) which consisted of all randomized participants who received at least 1 dose of study drug. In the FAS, participants were allocated to the treatment arm corresponding to the study medication that the participant was randomized to (treatment allocation as randomized).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 98 | 44
percentage of participants | 77.6 [68.0 to 85.4] | 70.5 [54.8 to 83.2]
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Adjusted difference of CCR at EOT + 2 Days. Adjusted treatment difference of proportions was calculated using a stratified Cochran-Mantel-Haenszel (CMH) method. Newcombe 95% confidence intervals (CIs) presented for adjusted treatment difference; Test type: Other; adjusted treatment difference = 7.5, 95% CI 2-sided [-7.4 to 23.9]

2. Secondary Outcome: Percentage of Participants With Sustained Clinical Response (SCR) at EOT +9 Days
Description: SCR at EOT + 9 days was defined as CCR (EOT + 2 days) without CDAD recurrence until assessment at EOT +9 days during the follow-up period. Recurrence for ages from birth to < 2 years was defined as re-establishment of watery diarrhea after CCR to an extent that was greater than that noted on the last day of study drug with positive direct or indirect testing for the presence of toxigenic Clostridium difficile (C. difficile) in stool and that, in the investigator's opinion, required retreatment with CDAD anti-infective therapy. Recurrence for ages ≥ 2 years < 18 years was defined as re-establishment of diarrhea after CCR to an extent (as measured by the frequency of UBMs) that was greater than that noted on the last day of study drug with positive direct or indirect testing for the presence of toxigenic C. difficile in stool and that, in the investigator's opinion, required retreatment with CDAD anti-infective therapy.
Time Frame: Up to day 19
Population: The analysis population consisted of the FAS (participants with CCR at EOT +2 days).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 76 | 31
percentage of participants | 94.7 [87.1 to 98.5] | 77.4 [58.9 to 90.4]
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Adjusted difference of SCR at EOT +9 days. Adjusted treatment difference of proportions was calculated using a stratified CMH method. Newcombe 95% CIs presented for adjusted treatment difference; Test type: Other; adjusted treatment difference = 16.3, 95% CI 2-sided [1.8 to 34.2]

3. Secondary Outcome: Percentage of Participants With Global Cure (GC) at EOT +9 Days
Description: GC was reported as a positive (Yes) or negative (No) outcome and was calculated using SCR and ICR/CCR values according to the following conditions: ● if ICR/CCR=Yes and SCR=Yes, then Global Cure was Yes. ● if ICR/CCR=Yes and SCR =No, then Global Cure was No. ● if ICR/CCR=No (SCR not assessed), then Global Cure was No. ● if ICR/CCR=Missing (SCR not assessed), then Global Cure was set to No. No multiple imputation method (MI) was used for global cure at EOT + 9 days.
Time Frame: Up to day 19
Population: The analysis population consisted of the FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 98 | 44
percentage of participants | 75.5 [65.8 to 83.6] | 54.5 [38.8 to 69.6]
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Adjusted difference of GC at EOT +9 days. Adjusted treatment difference of rates was calculated using a stratified CMH method. Newcombe 95% CIs presented for adjusted treatment difference; Test type: Other; adjusted treatment difference = 21.3, 95% CI 2-sided [4.5 to 37.7]

4. Secondary Outcome: Percentage of Participants With Recurrence of CDAD at EOT +9 Days
Description: Recurrence for ages from birth to < 2 years was defined as re-establishment of watery diarrhea after CCR to an extent that was greater than that noted on the last day of study drug with positive direct or indirect testing for the presence of toxigenic C. difficile in stool and that, in the investigator's opinion, required retreatment with CDAD anti-infective therapy. Recurrence for ages ≥ 2 years < 18 years was defined as re-establishment of diarrhea after CCR to an extent (as measured by the frequency of UBMs) that was greater than that noted on the last day of study drug with positive direct or indirect testing for the presence of toxigenic C. difficile in stool and that, in the investigator's opinion, required retreatment with CDAD anti-infective therapy.
Time Frame: Up to day 19
Population: The analysis population consisted of the FAS (participants with CCR at EOT +2 days).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 76 | 31
percentage of participants | 5.3 [1.5 to 12.9] | 22.6 [9.6 to 41.1]
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Adjusted difference of CDAD recurrence at EOT +9 days. Adjusted treatment difference of proportions was calculated using a stratified CMH method. Newcombe 95% CIs presented for adjusted treatment difference; Test type: Other; adjusted treatment difference = -16.3, 95% CI 2-sided [-34.2 to -1.8]

5. Secondary Outcome: Percentage of Participants With SCR at EOT +16 Days
Description: SCR at EOT + 16 days was defined as CCR (EOT + 2 days) without CDAD recurrence until assessment at EOT + 16 days during the follow-up period. Recurrence for ages from birth to < 2 years was defined as re-establishment of watery diarrhea after CCR to an extent that was greater than that noted on the last day of study drug with positive direct or indirect testing for the presence of toxigenic C. difficile in stool and that, in the investigator's opinion, required retreatment with CDAD anti-infective therapy. Recurrence for ages ≥ 2 years < 18 years was defined as re-establishment of diarrhea after CCR to an extent (as measured by the frequency of UBMs) that was greater than that noted on the last day of study drug with positive direct or indirect testing for the presence of toxigenic C. difficile in stool and that, in the investigator's opinion, required retreatment with CDAD anti-infective therapy.
Time Frame: Up to day 26
Population: The analysis population consisted of the FAS (participants with CCR at EOT +2 days).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 76 | 31
percentage of participants | 89.5 [80.3 to 95.3] | 71.0 [52.0 to 85.8]
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Adjusted difference of SCR at EOT +16 days. Adjusted treatment difference of proportions was calculated using a stratified CMH method. Newcombe 95% CIs presented for adjusted treatment difference; Test type: Other; adjusted treatment difference = 17.2, 95% CI 2-sided [1.9 to 35.6]

6. Secondary Outcome: Percentage of Participants With GC at EOT +16 Days
Description: GC was reported as a positive (Yes) or negative (No) outcome and was calculated using SCR and ICR/CCR values according to the following conditions: ● if ICR/CCR=Yes and SCR=Yes, then Global Cure was Yes. ● if ICR/CCR=Yes and SCR =No, then Global Cure was No. ● if ICR/CCR=No (SCR not assessed), then Global Cure was No. ● if ICR/CCR=Missing (SCR not assessed), then Global Cure was set to No. No multiple imputation method (MI) was used for global cure at EOT + 16 days.
Time Frame: Up to day 26
Population: The analysis population consisted of the FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 98 | 44
percentage of participants | 71.4 [61.4 to 80.1] | 52.3 [36.7 to 67.5]
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Adjusted difference of GC at EOT +16 days. Adjusted treatment difference of rates was calculated using a stratified CMH method. Newcombe 95% CIs presented for adjusted treatment difference; Test type: Other; adjusted treatment difference = 19.4, 95% CI 2-sided [2.3 to 35.9]

7. Secondary Outcome: Percentage of Participants With Recurrence of CDAD at EOT +16 Days
Description: as for outcome 4
Time Frame: Up to day 26
Population: The analysis population consisted of the FAS (participants with CCR at EOT +2 days).
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 76 | 31
percentage of participants | 7.9 [3.0 to 16.4] | 25.8 [11.9 to 44.6]
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Adjusted difference of CDAD Recurrence at EOT +16 days. Adjusted treatment difference of proportions was calculated using a stratified CMH method. Newcombe 95% CIs presented for adjusted treatment difference; Test type: Other; adjusted treatment difference = -17.2, 95% CI 2-sided [-35.6 to -1.9]

8. Secondary Outcome: Percentage of Participants With SCR at EOT +23 Days
Description: SCR at EOT + 23 days was defined as CCR (EOT + 2 days) without CDAD recurrence until assessment at EOT + 16 days during the follow-up period. Recurrence for ages from birth to < 2 years was defined as re-establishment of watery diarrhea after CCR to an extent that was greater than that noted on the last day of study drug with positive direct or indirect testing for the presence of toxigenic C. difficile in stool and that, in the investigator's opinion, required retreatment with CDAD anti-infective therapy. Recurrence for ages ≥ 2 years < 18 years was defined as re-establishment of diarrhea after CCR to an extent (as measured by the frequency of UBMs) that was greater than that noted on the last day of study drug with positive direct or indirect testing for the presence of toxigenic C. difficile in stool and that, in the investigator's opinion, required retreatment with CDAD anti-infective therapy.
Time Frame: Up to day 33
Population: The analysis population consisted of the FAS (participants with CCR at EOT +2 days).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 76 | 31
percentage of participants | 85.5 [75.6 to 92.5] | 71.0 [52.0 to 85.8]
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Adjusted difference of SCR at EOT +23 days. Adjusted treatment difference of proportions was calculated using a stratified CMH method. Newcombe 95% CIs presented for adjusted treatment difference; Test type: Other; adjusted treatment difference = 15.8, 95% CI 2-sided [-0.5 to 34.5]

9. Secondary Outcome: Percentage of Participants With GC at EOT +23 Days
Description: GC was reported as a positive (Yes) or negative (No) outcome and was calculated using SCR and ICR/CCR values according to the following conditions: ● if ICR/CCR=Yes and SCR=Yes, then Global Cure was Yes. ● if ICR/CCR=Yes and SCR =No, then Global Cure was No. ● if ICR/CCR=No (SCR not assessed), then Global Cure was No. ● if ICR/CCR=Missing (SCR not assessed), then Global Cure was set to No. No multiple imputation method (MI) was used for global cure at EOT + 23 days.
Time Frame: Up to day 33
Population: The analysis population consisted of the FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 98 | 44
percentage of participants | 68.4 [58.2 to 77.4] | 50.0 [34.6 to 65.4]
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Adjusted difference of GC at EOT +23 days. Adjusted treatment difference of rates was calculated using a stratified CMH method. Newcombe 95% CIs presented for adjusted treatment difference; Test type: Other; adjusted treatment difference = 18.8, 95% CI 2-sided [1.5 to 35.3]

10. Secondary Outcome: Percentage of Participants With Recurrence of CDAD at EOT +23 Days
Description: as for outcome 4
Time Frame: Up to day 33
Population: The analysis population consisted of the FAS (participants with CCR at EOT +2 days).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 76 | 31
percentage of participants | 11.8 [5.6 to 21.3] | 29.0 [14.2 to 48.0]
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Adjusted difference of CDAD Recurrence at EOT +23 days. Adjusted treatment difference of proportions was calculated using a stratified CMH method. Newcombe 95% CIs presented for adjusted treatment difference; Test type: Other; adjusted treatment difference = -15.8, 95% CI 2-sided [-34.5 to 0.5]

11. Secondary Outcome: Percentage of Participants With SCR at End of Study (EOS) (EOT +30 Days)
Description: SCR at EOS was defined as CCR (EOT + 2 days) without CDAD recurrence until assessment at EOS (EOT + 30 days) during the follow-up period. Recurrence for ages from birth to < 2 years was defined as re-establishment of watery diarrhea after CCR to an extent that was greater than that noted on the last day of study drug with positive direct or indirect testing for the presence of toxigenic C. difficile in stool and that, in the investigator's opinion, required retreatment with CDAD anti-infective therapy. Recurrence for ages ≥ 2 years < 18 years was defined as re-establishment of diarrhea after CCR to an extent (as measured by the frequency of UBMs) that was greater than that noted on the last day of study drug with positive direct or indirect testing for the presence of toxigenic C. difficile in stool and that, in the investigator's opinion, required retreatment with CDAD anti-infective therapy.
Time Frame: Up to day 40
Population: The analysis population consisted of the FAS (participants with CCR at EOT +2 days).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 76 | 31
percentage of participants | 85.5 [75.6 to 92.5] | 71.0 [52.0 to 85.8]
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Adjusted difference of SCR at EOS (EOT +30 days). Adjusted treatment difference of proportions was calculated using a stratified CMH method. Newcombe 95% CIs presented for adjusted treatment difference; Test type: Other; adjusted treatment difference = 15.8, 95% CI 2-sided [-0.5 to 34.5]

12. Secondary Outcome: Percentage of Participants With GC at EOS (EOT +30 Days)
Description: GC was reported as a positive (Yes) or negative (No) outcome and was calculated using SCR and ICR/CCR values according to the following conditions: ● if ICR/CCR=Yes and SCR=Yes, then Global Cure was Yes. ● if ICR/CCR=Yes and SCR =No, then Global Cure was No. ● if ICR/CCR=No (SCR not assessed), then Global Cure was No. ● if ICR/CCR=Missing (SCR not assessed), then Global Cure was set to No. Global Cure at EOT +30 days was derived using MI in case ICR/CCR=Missing (SCR not assessed) following Rubin's multiple imputation method.
Time Frame: Up to day 40
Population: The analysis population consisted of the FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 98 | 44
percentage of participants | 68.4 [58.2 to 77.4] | 50.0 [34.6 to 65.4]
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Adjusted difference of GC at EOS (EOT +30 days). Adjusted treatment difference of rates was calculated using a stratified CMH method. Newcombe 95% CIs presented for adjusted treatment difference; Test type: Other; adjusted treatment difference = 18.8, 95% CI 2-sided [1.5 to 35.3]

13. Secondary Outcome: Percentage of Participants With Recurrence of CDAD at EOS (EOT +30 Days)
Description: as for outcome 4
Time Frame: Up to day 40
Population: The analysis population consisted of the FAS (participants with CCR at EOT +2 days).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 76 | 31
percentage of participants | 11.8 [5.6 to 21.3] | 29.0 [14.2 to 48.0]
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Adjusted difference of CDAD recurrence at EOS/EOT +30 days. Adjusted treatment difference of proportions was calculated using a stratified CMH method. Newcombe 95% CIs presented for adjusted treatment difference; Test type: Other — Newcombe 95% CIs presented for adjusted treatment difference; adjusted treatment difference = -15.8, 95% CI 2-sided [-34.5 to 0.5]

14. Secondary Outcome: Time to Resolution of Diarrhea (TTROD)
Description: TTROD for ages from birth < 2 years was defined as time elapsing (hours rounded up from minutes > 30) from treatment start (time of first study drug dose) to diarrhea resolution (time of last episode of watery diarrhea the day prior to the first of 2 consecutive days without watery diarrhea sustained through EOT). TTROD for ages ≥ 2 years to < 18 years was defined as time elapsing (hours rounded up from minutes > 30) from treatment start (time of first dose) to diarrhea resolution (time of the last UBM the day prior to the first of 2 consecutive days of < 3 UBMs sustained through EOT). TTROD by Kaplan-Meier Method. Those who completed treatment but did not show diarrhea resolution until EOT were censored at Day 10/240 hours. Those who did not complete treatment, discontinued earlier but did not show diarrhea resolution until disc. day were censored at disc. (days converted to hours). Those whose diarrhea did not continue after first dose were included with a TTROD of 1 hour.
Time Frame: Up to day 10
Population: The analysis population consisted of the FAS.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 98 | 44
hours | 58 [29.0 to 122.0] | 97 [42.0 to 146.0]
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Time to resolution of diarrhea; Test type: Other; p = 0.579, Log Rank

15. Secondary Outcome: Time to Recurrence of CDAD for Participants With CCR at EOT +2 Days
Description: Time to recurrence was defined as the time (days) from CCR until the onset of recurrence. Time to recurrence of CDAD by Kaplan-Meier Method. Data for median was estimated and the 95% CI could not be estimated due to low event rate. Data not estimable denoted as NA. Participants with CCR at EOT+2 days, who completed the follow-up period but did not experience a recurrence of CDAD were censored at EOT+30 days and those who did not complete the follow-up period and discontinued during this period and did not experience a recurrence of CDAD were censored at day of discontinuation.
Time Frame: Up to day 40
Population: The analysis population consisted of the FAS (participants with CCR at EOT +2 days).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 76 | 31
days | 25 [NA to NA] — Data for Median was estimated and the 95% CI could not be estimated due to low event rate. | 26 [NA to NA] — Data for Median was estimated and the 95% CI could not be estimated due to low event rate.
Statistical Analysis 1: Comparison: Fidaxomicin vs Vancomycin; Time to recurrence of CDAD; Test type: Other; p = 0.023, Log Rank

16. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a study drug or who had undergone study procedures which did not necessarily have a causal relationship with this treatment. This included abnormal laboratory tests, vital signs, electrocardiogram data or physical examinations that were defined as AEs if the abnormality induced clinical signs or symptoms, required active intervention, interruption or discontinuation of study drug or was clinically significant in the investigator's opinion. The following standard with 3 grades was used to measure the severity of AEs, including abnormal clinical laboratory values: ● Mild: No disruption of normal daily activities ● Moderate: Affected normal daily activities ● Severe: Inability to perform daily activities. A treatment-emergent adverse event (TEAE) was defined as an AE observed after starting administration of the test drug/comparative drug.
Time Frame: From the first dose of study drug administration up to 30 days after EOT (up to day 40)
Population: The analysis population consisted of the safety analysis set (SAF), which consisted of all randomized participants who received at least 1 study drug dose. In the SAF, participants were allocated to the treatment arm corresponding to study drug first administered (fidaxomicin or vancomycin), even if it differed from the treatment randomized to.
Measure: Count of Participants; unit: Participants
Arm/Group | Fidaxomicin | Vancomycin
Number analyzed (Participants) | 98 | 44
Participants
  TEAE | 72 | 33
  Drug-related TEAE | 7 | 5
  Serious TEAE | 24 | 12
  Drug-related Serious TEAE | 0 | 0
  Moderate TEAE | 39 | 14
  Drug-related Moderate TEAE | 4 | 1
  Mild TEAE | 56 | 30
  Drug-related Mild TEAE | 3 | 4
  TEAE Leading to Death | 3 | 0
  Drug-related TEAE Leading to Death | 0 | 0
  TEAE leading to Withdrawal of Treatment (Tx) | 1 | 1
  Drug-related TEAE Leading to Withdrawal of Tx | 0 | 0

17. Secondary Outcome: Plasma Concentrations of Fidaxomicin
Description: Drug concentration was derived from the blood samples collected.
Time Frame: Within 30 minutes predose and 1 to 5 hours postdose taken between day 5 and day 10
Population: The analysis population consisted of the pharmacokinetics analysis set (PKAS). The PKAS consisted of all participants randomized to fidaxomicin, having received at least 1 dose of fidaxomicin and having at least 1 valid measurement of plasma concentration or fecal concentration of fidaxomicin or its main metabolite OP-1118.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Fidaxomin All Formulations: Participants received either fidaxomicin oral suspension or tablet formulation.
- Fidaxomicin Oral Suspension: Participants received fidaxomicin oral suspension formulation.
- Fidaxomicin Tablets: Participants received fidaxomicin tablets formulation.
Arm/Group | Fidaxomin All Formulations | Fidaxomicin Oral Suspension | Fidaxomicin Tablets
Number analyzed (Participants) | 98 | 67 | 31
ng/mL
  Predose: number analyzed (Participants) | 82 | 55 | 27
  Predose | 20.17 (40.16) | 15.26 (20.43) | 30.16 (63.27)
  Postdose: number analyzed (Participants) | 81 | 53 | 28
  Postdose | 39.41 (62.15) | 34.60 (57.79) | 48.53 (69.85)

18. Secondary Outcome: Plasma Concentrations of Metabolite OP-1118
Description: Drug concentration was derived from the blood samples collected.
Time Frame: Within 30 minutes predose and 1 to 5 hours postdose taken between day 5 and day 10
Population: The analysis population consisted of the PKAS.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fidaxomin All Formulations | Fidaxomicin Oral Suspension | Fidaxomicin Tablets
Number analyzed (Participants) | 98 | 67 | 31
ng/mL
  Predose: number analyzed (Participants) | 82 | 55 | 27
  Predose | 63.04 (171.97) | 42.18 (76.76) | 105.54 (277.67)
  Postdose: number analyzed (Participants) | 81 | 53 | 28
  Postdose | 116.64 (259.10) | 102.38 (245.19) | 143.63 (286.31)

19. Secondary Outcome: Metabolite-to-Parent Ratio (MPRconc)
Description: Drug concentration was derived from the blood samples collected.
Time Frame: Within 30 minutes predose and 1 to 5 hours postdose taken between day 5 and day 10
Population: The analysis population consisted of the PKAS.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Fidaxomin All Formulations | Fidaxomicin Oral Suspension | Fidaxomicin Tablets
Number analyzed (Participants) | 98 | 67 | 31
ratio
  Predose: number analyzed (Participants) | 82 | 55 | 27
  Predose | 3.18 (1.42) | 3.24 (1.46) | 3.05 (1.35)
  Postdose: number analyzed (Participants) | 81 | 53 | 28
  Postdose | 2.86 (1.18) | 2.95 (1.23) | 2.69 (1.06)

20. Secondary Outcome: Fecal Concentrations of Fidaxomicin
Description: Drug concentration was derived from the stool samples collected.
Time Frame: Within 24 hours of a dose taken between day 5 and day 10
Population: The analysis population consisted of the PKAS.
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Fidaxomin All Formulations | Fidaxomicin Oral Suspension | Fidaxomicin Tablets
Number analyzed (Participants) | 74 | 47 | 27
μg/g | 2685.56 (2476.92) | 2969.87 (2713.58) | 2190.63 (1948.68)

21. Secondary Outcome: Fecal Concentrations of Metabolite OP-1118
Description: Drug concentration was derived from the stool samples collected.
Time Frame: Within 24 hours of a dose taken between day 5 and day 10
Population: The analysis population consisted of the PKAS.
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Fidaxomin All Formulations | Fidaxomicin Oral Suspension | Fidaxomicin Tablets
Number analyzed (Participants) | 73 | 46 | 27
μg/g | 889.23 (817.83) | 789.15 (728.58) | 1059.73 (941.04)

22. Secondary Outcome: MPRconc Within 24 Hours of a Dose
Description: Drug concentration was derived from the stool samples collected.
Time Frame: Within 24 hours of a dose taken between day 5 and day 10
Population: The analysis population consisted of the PKAS.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Fidaxomin All Formulations | Fidaxomicin Oral Suspension | Fidaxomicin Tablets
Number analyzed (Participants) | 72 | 45 | 27
ratio | 0.43 (0.31) | 0.32 (0.19) | 0.63 (0.38)

23. Secondary Outcome: Acceptance of Formulation (Palatability Assessment) in All Participants at First Administration of Study Drug and at Day 7
Description: Acceptance of formulation was evaluated in all participants who received fidaxomicin oral suspension and vancomycin oral liquid (i.e., participants from birth to =< 6 years and participants > 6 years unable to swallow tablets) by means of a five-point rating scale (awful, poor, fair, good, excellent) by unblinded staff if hospitalized, and by the participant/parents/legal guardian when at home.
Time Frame: Days 1 and 7
Population: The analysis population consisted of the FAS.
Measure: Count of Participants; unit: Participants
Groups:
- Vancomycin Oral Liquid: Participants received vancomycin oral liquid formulation.
Arm/Group | Fidaxomicin Oral Suspension | Vancomycin Oral Liquid
Number analyzed (Participants) | 67 | 30
Participants
  Day 1 Awful | 4 | 5
  Day 1 Poor | 6 | 3
  Day 1 Fair | 13 | 6
  Day 1 Good | 19 | 7
  Day 1 Excellent | 13 | 4
  Day 1 Missing | 12 | 5
  Day 7 Awful | 2 | 3
  Day 7 Poor | 5 | 5
  Day 7 Fair | 8 | 5
  Day 7 Good | 21 | 9
  Day 7 Excellent | 16 | 3
  Day 7 Missing | 15 | 5

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration up to 30 days after EOT (up to day 40)
Description: The total number of deaths (all causes) includes deaths reported after time frame above.
Arm/Group | Fidaxomicin | Vancomycin
All-Cause Mortality (participants affected / at risk) | 3/98 | 2/44
Serious Adverse Events (participants affected / at risk) | 24/98 | 12/44
Other Adverse Events (participants affected / at risk) | 36/98 | 21/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fidaxomicin (N=98) | Vancomycin (N=44)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (6) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Mitochondrial encephalomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0)
Bacterial diarrhoea (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex meningoencephalitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Scedosporium infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Radiotherapy (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fidaxomicin (N=98) | Vancomycin (N=44)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 9 (11)
Constipation (Gastrointestinal disorders) | 5 (6) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 4 (5)
Vomiting (Gastrointestinal disorders) | 7 (8) | 6 (8)
Pyrexia (General disorders) | 11 (18) | 8 (11)
Oral candidiasis (Infections and infestations) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 8 (11) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2015-07-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT02218372/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT02218372/SAP_001.pdf